CLINICAL TRIAL: NCT00816062
Title: Endovascular Repair Using the Talent™ Abdominal Stent Graft System in Abdominal Aortic Aneurysms (VITALITY)
Brief Title: Post-Approval Trial of the Talent™ Abdominal Stent Graft to Treat Aortic Aneurysms
Acronym: VITALITY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiovascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P070027/S002
Record Dates: First submitted 2008-12-29; First posted 2008-12-31 (Estimated); Results first posted 2018-01-23 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Aortic Aneurysm, Abdominal
Keywords: Aortic Aneurysm; Aneurysm; Abdominal Aortic Aneurysm; Talent; Medtronic
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Aortic Aneurysm; Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): Patients diagnosed with an abdominal aortic or aorto-iliac aneurysm that are considered candidates for endovascular repair, per the FDA approved IFU.
  Interventions: Device: Talent Abdominal Stent Graft

INTERVENTIONS:
Device: Talent Abdominal Stent Graft — The Talent Abdominal Stent Graft is indicated for the endovascular treatment of abdominal aortic aneurysms with or without iliac involvement.

SUMMARY:
The purpose of this study is to examine, through the endpoints established in this protocol, the long-term safety and effectiveness of the Talent Abdominal Stent Graft System, in a post-approval environment.

DETAILED DESCRIPTION:
The Talent Abdominal Stent Graft System is a next-generation modular system for endovascular repair of Abdominal Aortic Aneurysm (AAA). The system was designed with the following enhancements: a suprarenal wire frame to provide migration resistance, and improved flexibility designed to treat difficult anatomies.

Medtronic Vascular submitted a Pre-Market Application (PMA) to the Food and Drug Administration (FDA) on October 17, 2007, and received market approval for the Talent Abdominal Stent Graft System on April 15th, 2008. As a condition of approval, the FDA has requested a post-approval study. Medtronic has therefore designed a post-approval study, in collaboration with FDA, to document the performance of the Talent Abdominal Stent Graft System under market conditions.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have an abdominal aortic aneurysm, with or without iliac involvement.
* Iliac/femoral access vessel morphology that is compatible with vascular access techniques, devices, and/or accessories;
* A proximal aortic neck length of ≥ 10mm;
* Proximal aortic neck angulation ≤ 60°;
* Distal iliac artery fixation length of ≥ 15mm;
* An aortic neck diameter of 18-32mm and iliac artery diameters of 8-22mm; and
* Vessel morphology suitable for endovascular repair.

Exclusion Criteria:

* Are less than 18 years of age
* Are pregnant or lactating
* Have a dominant patent inferior mesenteric artery and an occluded or stenotic celiac and/or superior mesenteric artery
* Have aneurysmal involvement or occlusion (surgically performed or naturally occurring) of the bilateral internal iliac arteries
* Have vessels and/or aneurysm dimensions that cannot accommodate the Talent Abdominal Stent Graft as per the indications in Section 3.
* Have no distal vascular bed (one vessel lower extremity run-off required)
* Have contraindications for use of contrast medium or anticoagulation drugs
* Have an uncorrectable coagulopathy
* Have an SVS/AAVS score greater than 2
* Have a mycotic aneurysm
* Have circumferential mural thrombus in the proximal aortic neck
* Have had a recent (within 3 months) myocardial infarction (MI), cerebral vascular accident (CVA), or major surgical intervention
* Have traumatic aortic injury
* Have leaking, pending rupture or ruptured aneurysms
* Have pseudoaneurysms resulting from previous graft placement
* Require a revision to previously placed endovascular stent grafts.
* Have genetic connective tissue disease (e.g., Marfan's or Ehlers-Danlos' Syndromes)
* Have concomitant thoracic aortic or thoracoabdominal aneurysms
* Are patients with active systemic infections
* Are patients who have a condition that threatens to infect the graft.
* Are patients with sensitivities or allergies to the device materials.
* Have access vessels (as determined by treating physician) that preclude safe insertion of the delivery system. NOTE: Iliac conduits may be used to ensure the safe insertion of the delivery system.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2008-12; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Luis Sanchez, MD, Principal Investigator — Washington University School of Medicine
Locations (18):
- United States (18):
  - USC Univerisity Hospital, Los Angeles, California
  - Palo Alto VAMC, Palo Alto, California
  - Christiana Care Health Services, Newark, Delaware
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - St. John's Medical Research Institute, Springfield, Missouri
  - Barnes Jewish, St Louis, Missouri
  - East Carolina University, Greenville, North Carolina
  - Forsyth Medical Center, Winston-Salem, North Carolina
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - Pinnacle Health Network, Harrisburg, Pennsylvania
  - Sanford USD Medical Center, Sioux Falls, South Dakota
  - North Central Heart Institute, Sioux Falls, South Dakota
  - St. Mary's Medical Center, Knoxville, Tennessee
  - Vanderbilt Vascular Surgery, Nashville, Tennessee
  - Wilford Hall Medical Center, Lackland Air Force Base, Texas
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Charleston Area Medical Center, Charleston, West Virginia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 166 subjects were enrolled in the previous cohort study (NCT # is not available). 94 subjects were enrolled into the Vitality study. When these two cohorts are combined it totals 260. The Vitality study collected information on its 94 enrolled subjects, but for study analysis both cohorts were combined.
Groups:
- Talent Abdominal Stent Graft: Patients diagnosed with an abdominal aortic or aorto-iliac aneurysm that are considered candidates for endovascular repair, per the Food and Drug Administration (FDA) approved Instructions for Use (IFU).
  >
  > Talent Abdominal Stent Graft: The Talent Abdominal Stent Graft is indicated for the endovascular treatment of abdominal aortic aneurysms with or without iliac involvement.
Period: Overall Study
Arm/Group | Talent Abdominal Stent Graft
Started | 260
Completed | 133
Not Completed | 127

BASELINE CHARACTERISTICS:
Groups:
- Treatment: Patients diagnosed with an abdominal aortic or aorto-iliac aneurysm that are considered candidates for endovascular repair, per the FDA approved IFU.>
  > Talent Abdominal Stent Graft: The Talent Abdominal Stent Graft is indicated for the endovascular treatment of abdominal aortic aneurysms with or without iliac involvement.
Arm/Group | Treatment
Number analyzed (Participants) | 260
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.7 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 227
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 254
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 241
  More than one race | 5
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 260

OUTCOME MEASURES:

1. Primary Outcome: Freedom From Aneurysm-related Mortality (ARM)
Description: ARM is defined as death from rupture of the abdominal aortic aneurysm or from any procedure intended to treat the Abdominal Aortic Aneurysm (AAA). If a death occurred within 30 days of any procedure intended to treat the AAA, then it is presumed to be aneurysm related unless there is evidence to the contrary. Deaths occurring after 30 days of any procedure intended to treat the AAA that are procedure-related should also be aneurysm related. All deaths were adjudicated by a Clinical Events Committee (CEC) to determine aneurysm, device and/or procedure relatedness.
Time Frame: 5 year Kaplan Meier (KM)
Population: All enrolled subjects.
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Treatment
Number analyzed (Participants) | 260
Proportion of participants | .97 [.946 to .994]

ADVERSE EVENTS:
Time Frame: 12 months
Groups:
- 1. Vitality: Medtronic Vitality
- 2. ELPS: Medtronic ELPS
Arm/Group | 1. Vitality | 2. ELPS
Serious Adverse Events (participants affected / at risk) | 31/94 | 99/166
Other Adverse Events (participants affected / at risk) | 5/94 | 112/166
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1. Vitality (N=94) | 2. ELPS (N=166)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 3 (3)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Heparin-Induced Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Angina Pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 3 (4) | 6 (6)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 2 (2)
Bradycardia (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac Failure (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac Failure Congestive (Cardiac disorders) | 4 (4) | 4 (4)
Cardiac Valve Disease (Cardiac disorders) | 0 (0) | 2 (3)
Cardiovascular Disorder (Cardiac disorders) | 0 (0) | 1 (1)
Coronary Artery Disease (Cardiac disorders) | 0 (0) | 3 (3)
Mitral Valve Incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 3 (3) | 3 (4)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal Distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal Ulcer Perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (2)
Inguinal Hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal Ischaemia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Intestinal Mass (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large Intestine Perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Retroperitoneal Fibrosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Catheter Site Pain (General disorders) | 0 (0) | 1 (1)
Chest Pain (General disorders) | 0 (0) | 3 (3)
Death (General disorders) | 0 (0) | 1 (1)
Device Deployment Issue (General disorders) | 0 (0) | 3 (3)
Device Dislocation (General disorders) | 0 (0) | 1 (1)
Device Kink (General disorders) | 0 (0) | 1 (1)
Hernia (General disorders) | 0 (0) | 1 (1)
Ill-Defined Disorder (General disorders) | 0 (0) | 4 (5)
Medical Device Complication (General disorders) | 0 (0) | 1 (1)
Oedema Peripheral (General disorders) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 2 (2) | 1 (1)
Stent Malfunction (General disorders) | 1 (1) | 0 (0)
Stent-Graft Endoleak (General disorders) | 2 (2) | 24 (32)
Hepatic Cyst (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic Lesion (Hepatobiliary disorders) | 0 (0) | 1 (1)
Candida Infection (Infections and infestations) | 0 (0) | 1 (1)
Groin Infection (Infections and infestations) | 0 (0) | 1 (1)
Incision Site Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 2 (2)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (2) | 0 (0)
Tracheobronchitis (Infections and infestations) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 2 (2)
Wound Infection (Infections and infestations) | 1 (1) | 0 (0)
Anaemia Postoperative (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Arterial Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Extradural Haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pelvic Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural Haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Seroma (Injury, poisoning and procedural complications) | 0 (0) | 5 (5)
Blood Creatinine Increased (Investigations) | 0 (0) | 3 (4)
Blood Glucose Increased (Investigations) | 0 (0) | 1 (1)
Catheterisation Cardiac (Investigations) | 0 (0) | 1 (1)
Haematocrit Decreased (Investigations) | 0 (0) | 2 (2)
Haemoglobin Decreased (Investigations) | 0 (0) | 2 (2)
Laboratory Test Abnormal (Investigations) | 0 (0) | 1 (1)
Platelet Count Decreased (Investigations) | 0 (0) | 1 (1)
Popliteal Pulse Increased (Investigations) | 0 (0) | 1 (1)
Red Blood Cell Analysis Abnormal (Investigations) | 0 (0) | 1 (1)
Urine Analysis Abnormal (Investigations) | 0 (0) | 1 (1)
Weight Increased (Investigations) | 0 (0) | 1 (1)
White Blood Cell Count Increased (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral Disc Degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle Tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adrenal Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bladder Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastrointestinal Stromal Tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Lung Squamous Cell Carcinoma Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Skin Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Throat Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Carotid Artery Stenosis (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular Accident (Nervous system disorders) | 1 (1) | 1 (1)
Dementia (Nervous system disorders) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Transient Ischaemic Attack (Nervous system disorders) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1)
Delirium Tremens (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Libido Decreased (Psychiatric disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 3 (3)
Renal Artery Occlusion (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal Disorder (Renal and urinary disorders) | 0 (0) | 4 (5)
Renal Failure (Renal and urinary disorders) | 3 (3) | 4 (4)
Renal Failure Chronic (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal Impairment (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal Infarct (Renal and urinary disorders) | 0 (0) | 2 (2)
Renal Ischaemia (Renal and urinary disorders) | 0 (0) | 1 (2)
Urinary Incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 1 (1) | 1 (1)
Genital Pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pelvic Fluid Collection (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Cardiac Pacemaker Insertion (Surgical and medical procedures) | 0 (0) | 1 (1)
Peripheral Artery Bypass (Surgical and medical procedures) | 0 (0) | 1 (1)
Renal Artery Angioplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
Ureteric Calculus Removal (Surgical and medical procedures) | 0 (0) | 1 (1)
Aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Aortic Aneurysm (Vascular disorders) | 1 (1) | 3 (3)
Aortic Dissection (Vascular disorders) | 1 (1) | 0 (0)
Aortic Stenosis (Vascular disorders) | 0 (0) | 1 (1)
Arterial Occlusive Disease (Vascular disorders) | 5 (5) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 2 (2)
Haemorrhage (Vascular disorders) | 0 (0) | 10 (10)
Hypotension (Vascular disorders) | 0 (0) | 3 (3)
Intermittent Claudication (Vascular disorders) | 0 (0) | 3 (3)
Peripheral Artery Dissection (Vascular disorders) | 1 (2) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Vascular Occlusion (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1. Vitality (N=94) | 2. ELPS (N=166)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 21 (24)
Ill-Defined Disorder (General disorders) | 0 (0) | 20 (31)
Pyrexia (General disorders) | 0 (0) | 21 (25)
Stent-Graft Endoleak (General disorders) | 5 (6) | 67 (146)
Seroma (Injury, poisoning and procedural complications) | 0 (0) | 15 (26)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 9 (9)
Renal Failure (Renal and urinary disorders) | 0 (0) | 9 (9)
Haemorrhage (Vascular disorders) | 0 (0) | 20 (22)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 60 days from the time submitted to the sponsor for review. The sponsor can require deletion of confidential information.The sponsor cannot require changes beyond those necessary to protect confidential information. The sponsor cannot extend the embargo.